CLINICAL TRIAL: NCT01361971
Title: Hyperbaric Oxygen Treatment Ameliorates Insulin Resistance
Acronym: HOTAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, A/Prof, University of Adelaide
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAH100615
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Insulin resistance; Inflammation; Hypoxia
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Treatment — Participants will undergo 4 treatments of hyperbaric oxygen. Each treatment consists of 90 minutes compression at 2 atmospheres of pressure, with 30 minutes decompression back to 1 atmosphere, during this time, patients will be treated with 100% Oxygen delivered via a hood system.

SUMMARY:
Obesity is an epidemic in Western society and is the biggest risk factor for insulin resistance and type 2 diabetes. The investigators have preliminary evidence showing that hyperbaric oxygen therapy rapidly increases insulin sensitivity in humans. This requires confirmation in a larger population, and with this study the investigators will also test for mechanisms how this occurs. The investigators suspect that modulation of hypoxia and stress response proteins following changes in tissue oxygenation may contribute to these improvements. This study has the potential to yield new and important insights into the insulin resistance in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese men with and without type 2 diabetes aged 45-70
* Lean men without type 2 diabetes aged 45-70

Exclusion Criteria:

* smokers
* claustrophobic
* sleep apnoea
* blood donor
* exercise more than 2 times per week
* under certain medications eg: bleomycin,corticosteroid

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 1 year
  Using Hyperinsulinemic clamp

SECONDARY OUTCOMES:
Hypoxia and inflammatory markers | 1 year
  using IHC, qPCR, Western blot

CONTACTS AND LOCATIONS:
Overall Officials: Leonie K Heilbronn, Phd, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia